CLINICAL TRIAL: NCT02827825
Title: Patients Undergoing Strokes Admitted in Intensive Care Requiring Neurosurgical ICU Crossing: Patient Profile and Prognosis
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AVC REANIMATION
Record Dates: First submitted 2016-06-30; First posted 2016-07-11 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2016-06

CONDITIONS: Cerebral Stroke
Keywords: Neurosurgical; Intensive Care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — No intervention. It's a study on retrospective Data

SUMMARY:
The aim of this study is to describe the population of patients admitted to the ICU in neurosurgery for stroke requiring secondary care in intensive care and their future.

DETAILED DESCRIPTION:
Methodology :

DESIGN:

Retrospective observational study single center, non-interventional Term study over 2 years, retrospectively

Acquisition of data:

* Study of computer file: report available on DxCare hospital and Cora
* Collection of data as excel spreadsheet
* Statistical analysis: local management
* Anonymity of data:

  * For each subject will be awarded an identifier (original name and surname - year of birth) and the data will be entered on a computer file which will be sent to the statistician in charge of analyzing the GHPSJ site. There will be no exchange of personal data for this study is single center on the site GHPSJ.

Development of the study:

* Procedure:

  * Series includable patients from the PMSI data
  * Select folders according the inclusion criteria
  * Collecting information from files on Excel spreadsheet by the internal charge of data collection (Sylvain CHAWKI)
  * Statistical Analysis
  * Writing Article
* Expected duration of patient recruitment: Retrospective of 2 and a half years from January 1, 2013 to April 31, 2015

ELIGIBILITY:
Inclusion Criteria:

* Admitted USINV for ischemic or hemorrhagic stroke
* Admitted secondarily in ICU

Exclusion Criteria:

* Admission in ICU in first
* Administrative Admission in Intensive Care Requiring Neurosurgical within the thrombolysis alert regulated by the neurovascular guard but going directly to ICU imaging waning
* Subarachnoid hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in Intensive Care Requiring Neurosurgical for ischemic or hemorrhagic stroke. then, admitted secondarily in ICU
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Death event | Day 1 after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: ZUBER Mathieru, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France